CLINICAL TRIAL: NCT04420442
Title: Influence of Surgical Scar Resection, Followed by Reconstruction With Integra and Split Skin Grafts on Quality of Life, Body Perception, Scar Perception and Stigmatization in Patients With Non-Suicidal Self-Inflicted Scars
Brief Title: Scar Resection and Reconstruction With Integra and Split Skin Grafts in Patients With Non-Suicidal Self-Inflicted Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Berufsgenossenschaftliche Unfallklinik Ludwigshafen (Other)
Collaborators: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Dimitra Kotsougiani-Fischer, Privat Dozent Doctor med., Berufsgenossenschaftliche Unfallklinik Ludwigshafen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BULudwigshafen
Record Dates: First submitted 2020-02-26; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Nonsuicidal Self Injury; Stigmatization; Cicatrix; Skin Transplantations
MeSH Terms: conditions — Self-Injurious Behavior; Stereotyping; Cicatrix | interventions — integra artificial skin

STUDY DESIGN:
Intervention Model Description: In this prospective monocentric non-randomized trial the intervention group and the control will be compared to each other. Furthermore, within the intervention group an intra-individual comparison will be carried out over the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Group (Active Comparator): In addition to the comparison between arm 1 and 2, there will be an intraindividual comparison within arm 1.
  Interventions: Procedure: Scar Transformation Group
- Control Group (No Intervention): No Intervention.

INTERVENTIONS:
Procedure: Scar Transformation Group — Surgical excision of the NSSI scars followed by IntegraTM transplantation and wound closure with a negative pressure wound system. After 21 days the silicone layer of the IntegraTM will be removed and split thickness skin will be transplanted. After suture removal a compression therapy by individually tailored garments will be started for 12 months.
  Other Names: Integra
  Arms: Intervention Group

SUMMARY:
Non-suicidal self-inflicted (NSSI) scars can act as a physical reminder of previous self-inflicted self-harm, thereby not only worsening the symptoms of depression and self-doubt but also leading to recurrent self-infliction and social exclusion. Several different treatment options exist to alter the appearance of NSSI scars like pulsed-dye laser therapy (PDL), non-ablative fractional laser therapy, dermabrasion or elliptical excision. However, none of these treatment options can completely diminish the scars. In the majority of cases, the unique scar pattern of NSSI scars and in addition to that the "reminder" remains. In contrast to regular scar revisions, the aesthetical appearance is not the most important outcome parameter as the main focus of the surgical treatment is destigmatization. The surgical transformation of the scar into a burn-like scar could change the scar-perception of the society and the patient, thereby improving the patient's quality of life and body perception. Surgical resection with preservation of the subcutaneous tissue followed by consecutive reconstruction with a bilayer dermal regenerative matrix (IntegraTM) and split skin grafts might represent a promising and novel therapeutic approach. The hypothesis is that by surgically transforming the non-suicidal self-inflicted scars into a burn-like scar the patient's body and scar perception will be positively altered and the stigmatization by the society reduced.

DETAILED DESCRIPTION:
Non-suicidal self-injury behaviour describes behaviour in patients, who have no intention to commit suicide. This can be performed in many different ways, e.g., automutilation through burning, scratching, or hitting. Often this behaviour results in deep scars and disfigurements. The prevalence of patients with NSSI scars is estimated to be 13.4% in adolescents and 5.5% in adults. Non-suicidal behaviour is often associated with other psychological diseases like personality disorders, character disorders of the Borderline type, anxiety, and substance abuse disorders. In these cases, usually, interdisciplinary therapy concepts are needed. A major problem is that the scars due to its constant confrontation can induce repetitive non-suicidal self-injury behaviour. Furthermore, the image of the NSSI scars leads to stigmatization by society and in addition to that to a withdrawal from society by the patients. Hence, the need for adequate treatment of the NSSI scars to relief the burden of stigmatization for the patients is immense. At the moment, non-invasive therapies like pulsed-dye laser therapy (PDL) and non-ablative fractional laser therapy, as well as minimal-invasive therapies like dermabrasion or elliptical excision offer one possible option, but the undoubted cause of the scar remains visible. At the moment only case studies exist which describe the beneficial effect of surgical resection followed by consecutive reconstruction with a dermal regenerative matrix and split skin grafts. These studies have evaluated the aesthetic outcome and briefly assessed the well-being of the patients. However, currently, no study exists investigating the effect of the two-step surgical procedure on body perception and the psychological outcome in general. The overall goal of the described study is to establish a therapy concept for patients who suffer from constant confrontation with their NSSI scars. Stigmatization by the society and by the patients themselves, body perception, quality of life, and scar perception will be evaluated over the study period of 36 months. Furthermore, the scar itself will be assessed using a cutometer and the scar image will be evaluated using the Patient and Observer Scar Assessment Scale.

The data analyses will be performed with SPSS, version 20.0, SPSS Inc. Chicago, USA. For the normally distributed values, the paired T-test will be used. Not normally distributed values will be analysed by the Wilcoxon signed-rank Test. The significance level will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-suicidal self-inflicted scars (NSSI) on the forearms who have resigned from self-infliction for more than one year can be included in the study.
* The patients have to be older than 18 years old. Their psychological status has to be stable and certified by a psychologist.
* Patients have to have a high psychosocial pressure due to the non-suicidal self-inflicted scars on the forearms.
* Patients have to agree to supportive psychotherapy during the time of the study.
* Patients have to agree to wear their compression gear for 12 months after the surgical intervention.

Exclusion Criteria:

* Pregnancies
* Age younger than 18
* Any other comorbid conditions like body-dysmorphic conditions or eating disorders
* Tendency to develop hypertrophic scars or keloids
* The participation in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
body perception - Multidimensional Body Self Relations AS Questionnaire | 36 months
  This questionnaire consists of 34 items that consists of 5 subscales. The items are rated on a 5 point likert scale. High scores indicate an increased dissatisfaction with body appearance and low scores indicate satisfaction with the body appearance. MBSRQ-AS subscale scores are the means of the constituent items after reversing contra-indicative items (i.e., 1 = 5, 2 = 4, 4 = 2, 5 = 1).
scar perception - Patient and Observer Scar Assessment Scale | 36 months
  The questionnaire consists of two scales (patient and observer scale) and each scale consists of 6 items. The maximum value is 60 (worst outcome) and the minimum value is 6 (best outcome). (POSAS).
quality of life: SF-36 questionnaire | 36 months
  This questionnaire consists of 36 items. The maximum value is 100 (best outcome) and the minimum value is 0 (worst outcome).
scar perception- Questionnaire for the evaluation of scar perception after burn trauma (FKBB) | 36 months
  The questionnaire consists of 23 items and three introduction questions. The maximum score of each item is 5 (good body perception) and the lowest score is 1 (bad body perception). The overall score is calculated through the mean of the whole scale. The three introduction questions have a score of 0 (bad body perception) and 10 (good body perception). The questions are not part of the overall result, they are needed for the overall body acceptance and thereby for calculating the correlation between body perception and acceptance.
stigmatization - Self Disgust Scale | 36 months
  The questionnaire is an 18-item scale. The items are rated on a 7-point likert scale. The maximum score was 84 and the minimum score was 12. A high score indicated high self-disgust and a low score indicated low self-disgust.
stigmatization - Self Regret Scale | 36 months
  The questionnaire is a 21-item scale. The items are rated on a 5-point likert scale. The maximum score was 105 and the minimum score was 21. A high score indicated high levels of regret and a low score indicated a low regret level.
stigmatization - Self-Stigma of Mental Illness Scale (SSMIS-SF) | 36 months
  This Scale consists of 4 subscales, each consisting of 5 items. On each subscale the maximum score is 45. There is no total score for the 4 subscales. The maximum score of each subscale is 45 and the minimum scale is 5. Higher scores are associated with higher levels of stigmatization.
stigmatization - Stigma Stress Scale | 36 months
  This scale consists of two subscales. Each subscale consists of 4 items. The maximum score of each subscale is 28 and the minimum score is 4. The first subscale analyses the perceived stigma-related harm and the second subscale analyses the perceived coping resources. For analyzing the level of stigma stress the difference between the two subscales is calculated (harm minus coping - from -6 to +6). Higher scores are associated with higher levels of stigma stress.
stigmatization - Disclosure of psychological illness in public and private surroundings - scale | 36 months
  Two items per subject. Highest score is 7 and the lowest score is 1. A low score indicates low levels of confidence with the patients psychological illness, whereby high scores indicate high levels of confidence with the psychological illness.
stigmatization - Internalized stigma of mental illness inventor (ISMII ) | 36 months
  This questionnaire consists of 5 items. The mean value is between 1 and 4. A high value is associated with a higher level of discrimination.
stigmatization - Self-labeling and Shame Scale | 36 months
  Two items per subject. Highest score is 9 and associated with a high level of self-labelling and shame. Lowest score is is one and associated with a low level of self-labelling and shame.

SECONDARY OUTCOMES:
scar image | 36 months
  An objective analysis of the image of the scar and its constitution will be performed with the use of a 3D camera and cutometer measurements. With the cutometer the skin elasticity can objectively be assessed.
satisfaction with the aesthetic appearance: non-validated subjective questionnaire | 36 months
  A non-validated subjective questionnaire, especially designed for the study with focus on the aesthetic satisfaction with the scar, will be used. The questionnaire will use likert scales (score 0-4) with the best-achievable score of 4 points reflecting the highest satisfaction with the reconstructive result.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitra Kotsougiani-Fischer, MD, Principal Investigator — Senior; Ulrich Kneser, MD, Study Chair — chief of department; Julian Vogelpohl, MD, Principal Investigator — Senior
Locations (1):
- BG Trauma Center Ludwigshafen, Ludwigshafen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Turner BJ, Austin SB, Chapman AL. Treating nonsuicidal self-injury: a systematic review of psychological and pharmacological interventions. Can J Psychiatry. 2014 Nov;59(11):576-85. doi: 10.1177/070674371405901103. PMID 25565473
- [Result] Swannell SV, Martin GE, Page A, Hasking P, St John NJ. Prevalence of nonsuicidal self-injury in nonclinical samples: systematic review, meta-analysis and meta-regression. Suicide Life Threat Behav. 2014 Jun;44(3):273-303. doi: 10.1111/sltb.12070. Epub 2014 Jan 15. PMID 24422986
- [Result] Nitkowski D, Petermann F. [Non-suicidal self-injury and comorbid mental disorders: a review]. Fortschr Neurol Psychiatr. 2011 Jan;79(1):9-20. doi: 10.1055/s-0029-1245772. Epub 2010 Nov 22. German. PMID 21104583
- [Result] Monstrey S, Middelkoop E, Vranckx JJ, Bassetto F, Ziegler UE, Meaume S, Teot L. Updated scar management practical guidelines: non-invasive and invasive measures. J Plast Reconstr Aesthet Surg. 2014 Aug;67(8):1017-25. doi: 10.1016/j.bjps.2014.04.011. Epub 2014 May 14. PMID 24888226
- [Result] Chou CY, Chang HA, Chiao HY, Wang CY, Sun YS, Chen SG, Wang CH. Interchangeable skin grafting to camouflage self-inflicted wound scars on the dorsal and volar forearm: a case report. Ostomy Wound Manage. 2014 Apr;60(4):50-2. PMID 24706403
- [Result] Bachtelle SE, Pepper CM. The Physical Results of Nonsuicidal Self-Injury: The Meaning Behind the Scars. J Nerv Ment Dis. 2015 Dec;203(12):927-933. doi: 10.1097/NMD.0000000000000398. PMID 26524516